CLINICAL TRIAL: NCT02175667
Title: Influence of the Global Postural Reeducation and the Personality Traits in the Range of Motion, in the Stabilometry and in the Postural Sway.
Brief Title: Influence of the Global Postural Reeducation and the Personality in the Posture
Acronym: RPG-POSTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Carlos Lozano Quijada, PT, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DPC-CLQ-001-12
Record Dates: First submitted 2014-06-16; First posted 2014-06-26 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2014-10

CONDITIONS: Postural; Defect
Keywords: Global postural reeducation; Stabilometry; Postural Sway; Range of motion; Personality traits
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Global Postural Reeducation (Experimental): Participants receiving GPR treatment during 45 minutes to stretch muscular chains
  Interventions: Procedure: Global Postural Reeducation
- Control (No Intervention): Participants not receiving GPR treatment

INTERVENTIONS:
Procedure: Global Postural Reeducation — Experimental group is treated in a 45 minutes GPR session, with three postures: the first was for the anterior muscular chain with the patient lying supine on a couch with arms at 45 degrees, hips open, and feet in opposition on top of the table. This posture is maintained 25-30 minutes. The second GPR posture, to stretch the posterior muscle chain, the participant is positioned with legs elevated, for 12-15 minutes. Third position is with the participant standing and 2-5 minutes to integrate the postural corrections. During all the time, the physiotherapist use manual therapy for stretch the muscles under the official rules of GPR techniques. Group control do not receive any technique.
  Other Names: Manual Therapy; Muscle chains; Stretching
  Arms: Global Postural Reeducation

SUMMARY:
Determine the influence of a treatment with Global Postural Reeducation techniques and the personality traits in the stabilometric parameters

DETAILED DESCRIPTION:
This study is realized with university students. For a first objective of this study, all the participants complete the "big five questionnaire" to determine their personality traits and then the subjects are analyzed with a stabilometric platform and cervical/lumbar range of motion (ROM) to determine their basal parameters. The personality traits and the basal stabilometric parameters like the postural sway, will be crossed to investigate a possible relation. For a second objective, the randomized study of the effectiveness of the Global Postural Reeducation (GPR) in the stabilometric parameters, the subjects are divided in a experimental group or in a control group. Experimental group is treated in a 45 minutes GPR session, with three postures: the first is for stretch the anterior muscular chain with the patient lying supine on a couch with arms at 45 degrees, hips open, and feet in opposition on top of the couch. This posture is maintained 25-30 minutes. In the second GPR posture, to stretch the posterior muscular chain, the subject is positioned with legs elevated, for 12-15 minutes. Third position is with the participant in upright standing posture 2-5 minutes to integrate the postural corrections. During all the time, the physiotherapist uses manual therapy for stretch the muscles under the official rules of GPR techniques. Group control do not receive any technique. After the time of the intervention or no intervention, a second measure of stabilometric parameters and ROM is taken. After this first day, two days later and seven days later, the measures are repeated to determinate the permanence of the effects of GPR techniques.

The improvement will be assessed by calculating indicators of clinical relevance: relative risk (RR), absolute risk reduction (AR). The results will be compared statistically to determine some possible relation. The confidence intervals (CI) will be calculated for the most relevant parameters. The analysis will be made with a statistics program (SPSS 19.0)

ELIGIBILITY:
Inclusion Criteria:

* College students spend 4 hours or more per day sitting

Exclusion Criteria:

* College students do not spend 4 hours or more per day sitting.
* Subjects with a traumatic problem, injuries, in the moment of the study, or subject in treatment of this injuries

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Centre of pressure displacement in standing position | Before intervention, 2 minutes after, 2 days after, 7 days after
  Displacement antero-posterior and lateral of COP measured with a platform of pressures

SECONDARY OUTCOMES:
Plantar pressures distribution in standing position | Before intervention, 2 minutes after, 2 days after, 7 days after
  Plantar pressures distribution in each foot measured with a platform of pressures
Percentage of load distribution in standing position | Before intervention, 2 minutes after, 2 days after, 7 days after
  Load distribution between feet measured with a platform of pressures
Lumbar and cervical range of motion | Before intervention, 10 minutes after, 2 days after, 7 days after
  Cervical and lumbar inclinometer for goniometry

OTHER OUTCOMES:
Big Five personality traits questionnaire (spanish version) | Before intervention
  Auto-reported questionnaire for individual score in the five broad dimensions of personality: openness to experience, conscientiousness, extraversion, agreeableness, and neuroticism.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Lozano-Quijada, PT, Principal Investigator — Universidad Miguel Hernández; Emilio J Poveda-Pagán, PhD, Study Director — Universidad Miguel Hernandez de Elche; María J Prieto-Castelló, PhD, Study Director — Universidad Miguel Hernández
Locations (1):
- Miguel Hernández University of Elche, Sant Joan, Alicante, Spain